CLINICAL TRIAL: NCT03053076
Title: Safety and Efficacy of Autologous Umbilical Cord Blood Mononuclear Cells Transfusion in Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, Professor, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GuangdongWCH
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Safety Issues; Effect of Drugs; Neonatal Death
Keywords: cord blood mononuclear cells; safety; effect; neonates
MeSH Terms: conditions — Perinatal Death | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo1 (Placebo Comparator): 0.9% sodium chloride infusion 48 hours after birth ,the infusion speed is 4ml/kg/h， 8-12h，
  Interventions: Drug: 0.9% Sodium Chloride
- CBMNC (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells Therapy 48 hours after birth ,dose is 25 million cells/kg ，the infusion speed is 4ml/kg/h， 8-12h，
  Interventions: Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy

INTERVENTIONS:
Other: Autologous Umbilical Cord Blood Mononuclear Cells Therapy — Autologous Umbilical Cord Blood Mononuclear Cells Therapy in preterm for safety and effect evaluation
  Arms: CBMNC
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride in control group
  Arms: Placebo1

SUMMARY:
To study the safety and efficacy of Autologous Umbilical Cord Blood Mononuclear Cells transfusion on clinical outcome in preterm infants

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial that constitutes two time points cohorts with 100 participants per cohort who will receive intravenous doses of Autologous Umbilical Cord Blood Mononuclear Cells --25 million cells/kg, 48 hours after birth. And the placebo will be 0.9% sodium chloride.The investigator will proceed the groups during the same period.

1. Demographic Data and Baseline Characteristics of the Studied Groups were collected:

   * Gestational age (weeks)
   * Birth weight (g)
   * gender
   * Cesarean section delivery
   * Antenatal steroids
   * Prolonged rupture of membrane
   * Multiple pregnancies
   * APGAR score at 5 minutes
   * Thrombocytopenia before intervention
   * CRP before intervention (mg/L)
   * TNF-α(tumor necrosis factor α ) before intervention (pg/mL)
2. Assessment of clinical condition in the course by measurement of arterial blood pressure, heart and respiratory rates and skin temperature was recorded continuously
3. Autologous cord blood mononuclear cells doses is 25 million cells/kg ，the infusion speed is 4ml/kg/h， 8-12h，and with same volume of 0.9% sodium chloride as placebo.
4. The following are monitored at 3、7、14、21 days after birth:

   * mortality, incidence of sepsis, neonatal respiratory distress syndrome (NRDS), bronchopulmonary dysplasia (BPD), retinopathy of prematurity (ROP), necrotising enterocolitis (NEC), intraventricular haemorrhage (IVH), Hypoxic Ischemic Encephalopathy (HIE), anaemia, thrombocytopenia, neutrophil,TBNK cells subgroup, before hospital discharge.
5. Long-term follow up: in 1m, 3m, 6m,1y: neurodevelopment [Bayley Scales of Infant], asthma, anemia and physique growth.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-eight weeks to thirty-seven weeks

Exclusion Criteria:

* Preterm infants with major congenital malformations, chromosomal anomalies, inborn errors of metabolism and clinical or laboratory evidence of a congenital infection

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-05-15 (Estimated); Study Completion 2017-05-15 (Estimated)

PRIMARY OUTCOMES:
number of patients who died | up tp 21 days after birth
  mortality rate

SECONDARY OUTCOMES:
number of patients with neurodevelopmental disorder assessed by Bayley Score | up to 1 month, 3 months, 6 months and 1 year
  Long term follow up: in 1 month, 3 months, 6 months, and 1 year: neuro-development

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, Phd, Principal Investigator — Guangdong Women and Children Hospital
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ballen KK, Gluckman E, Broxmeyer HE. Umbilical cord blood transplantation: the first 25 years and beyond. Blood. 2013 Jul 25;122(4):491-8. doi: 10.1182/blood-2013-02-453175. Epub 2013 May 14. PMID 23673863
- [Derived] Ren Z, Fang X, Zhang Q, Mai YG, Tang XY, Wang QQ, Lai CH, Mo WH, Dai YH, Meng Q, Wu J, Ao ZZ, Jiang HQ, Yang Y, Qu LH, Deng CB, Wei W, Li Y, Wang QI, Yang J. Use of Autologous Cord Blood Mononuclear Cells Infusion for the Prevention of Bronchopulmonary Dysplasia in Extremely Preterm Neonates: A Study Protocol for a Placebo-Controlled Randomized Multicenter Trial [NCT03053076]. Front Pediatr. 2020 Apr 2;8:136. doi: 10.3389/fped.2020.00136. eCollection 2020. PMID 32300579